CLINICAL TRIAL: NCT04176705
Title: Pilot Study of Early Postoperative Fractional Ablative Laser Treatment of Skin Grafts for Burns
Brief Title: Fractional Ablative Laser Treatment for Skin Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00058363
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2023-07

CONDITIONS: Burn Scar; Skin Graft Scar
Keywords: Fractional laser; Ablative Laser; Carbon Dioxide Laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Laser (Experimental): Split person design. Each participant had a skin burn area that was treated with the laser and a skin burn area that was not treated with the laser.
  Interventions: Drug: Lidocaine Cream; Drug: Triamcinolone Acetonide Cream; Device: Fractional Ablative Laser
- No laser (Placebo Comparator): Split person design. Each participant had a skin burn area that was treated with the laser and a skin burn area that was not treated with the laser.
  Interventions: Drug: Lidocaine Cream; Drug: Triamcinolone Acetonide Cream

INTERVENTIONS:
Drug: Lidocaine Cream — Both sites will have lidocaine 4% topical anesthetic cream (Ferndale Laboratories, Ferndale MI) applied as thin layer and left for 30-45 minutes to minimize discomfort applied before laser treatment.
Drug: Triamcinolone Acetonide Cream — Triamcinolone acetonide cream (Bristol-Myers Squibb, Princeton, NJ) at a concentration of 20mg/ml will be applied immediately after treatment to both laser and no-laser sites - as this is often reported and there is some speculation that this may be part of the reason improvement is noted.
Device: Fractional Ablative Laser — Applied to only site that is randomized to laser intervention
  Arms: Laser

SUMMARY:
Doctors and patients refer to all areas of skin changes from burn injury as burn scars. However, different areas of scars from burns can be treated differently. The burn scars that come from skin grafting surgery might be improved with laser treatment. The purpose of this study is to see if treating burn skin graft scars with a laser could make it better.

Fractional Ablative Laser has been approved by the US Food and Drug Administration (FDA), but it has not been approved for use in the early stages of scar maturation and is considered investigational for this study.

DETAILED DESCRIPTION:
This pilot study is being conducted to establish safety, however the study team will make multiple measures to measure for efficacy as well. The study team hypothesizes that human split-thickness skin grafts will safely respond similar to the porcine model when treated with the Fractional Carbon Dioxide (FxCO2) laser and have significantly less secondary contracture than control sites. The great majority of laser studies have addressed treatment of established scars. Ideally, treatment modalities could be moved into the acute period of injury, to shorten the recovery time of thermal burns by decreasing the time to maximum recovery, and mitigate scar formation. The current study will address the impact on treatment of skin graft applied in the treatment of acute burn wounds. Preliminary work completed by our team has confirmed that the red Duroc porcine model is a good model of hypertrophic scar formation in humans, and early use of the FxCO2 on split-thickness skin grafts decreased secondary contracture. Further, the study team has identified a period of 19 weeks between the time custom-made compression garments are ordered and actually applied with benefit to the patient. The study team has identified a "therapeutic donut hole" in which they have no efficacious alternative to offer until about 19 weeks. In these patients who had larger burn returning to the OR for additional procedures, the study team was able to offer FxCO2 treatment as a "salvage" therapy. With this, the study team has demonstrated safety for the skin graft and anecdotal efficacy. The study team proposes a pilot study to prospectively demonstrate safety in a controlled study and attempt to establish efficacy of early (post grafting day 7-10) FxCO2 laser treatment of split-thickness skin graft applied in the treatment of burn injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are to undergo skin grafting procedures for acute treatment of thermal burns.
* Patients with grafts placed over at least 100cm^2

Exclusion Criteria:

* Patients who have are not scheduled to undergo skin grafting procedures
* Patients who have grafts placed under 100cm^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Bailey, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We will plan to share individual participant data with other researchers. We welcome critical examination of the protocol, statistical analysis of recorded data, informed consent form, and clinical study report. We are happy to share de-identified data (original photo files, tracings, and recorded measures of skin quality) and responses to questionnaires.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available within 6 months of data completion.
Access Criteria: Research groups with authors who have at least one related publication

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each of the nine subjects had two burned areas. One area was treated with laser and the other area was not treated.
Units Other Than Participants: skin burn areas
Period: Overall Study
Arm/Group | Laser | No Laser
Started | 9; 9 skin burn areas | 9; 9 skin burn areas
Completed | 1; 1 skin burn areas | 1; 1 skin burn areas
Not Completed | 8; 8 skin burn areas | 8; 8 skin burn areas
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Population: A total of nine subjects were enrolled. Each of the nine subjects had two burned areas. Each had one area treated with laser and the other area was not treated.
Groups:
- Overall Participants: This is a split person design. Overall participants in both arms are included here.
Arm/Group | Overall Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Contracture of Scar Surface Area (Percentage of Original Area)
Description: Contracture of Scar Surface Area 90 days post grafting: The surface area of the skin graft cm^2 at about 90 days after skin grafting will be compared to the size of the original skin graft at about one week after surgery.
Time Frame: 90 days post-grafting
Population: One subject withdrew after signing consent.
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: skin burn area
Groups:
- Laser: Split person design.
  Lidocaine Cream: Both sites will have lidocaine 4% topical anesthetic cream (Ferndale Laboratories, Ferndale MI) applied as thin layer and left for 30-45 minutes to minimize discomfort applied before laser treatment.
  Triamcinolone Acetonide Cream: Triamcinolone acetonide cream (Bristol-Myers Squibb, Princeton, NJ) at a concentration of 20mg/ml will be applied immediately after treatment to both laser and no-laser sites - as this is often reported and there is some speculation that this may be part of the reason improvement is noted.
  Fractional Ablative Laser: Applied to only site that is randomized to laser intervention
- No Laser: Split person design.
  Lidocaine Cream: Both sites will have lidocaine 4% topical anesthetic cream (Ferndale Laboratories, Ferndale MI) applied as thin layer and left for 30-45 minutes to minimize discomfort applied before laser treatment.
  Triamcinolone Acetonide Cream: Triamcinolone acetonide cream (Bristol-Myers Squibb, Princeton, NJ) at a concentration of 20mg/ml will be applied immediately after treatment to both laser and no-laser sites - as this is often reported and there is some speculation that this may be part of the reason improvement is noted.
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 8 | 8
Number analyzed (skin burn area) | 8 | 8
percentage | 97 (14) | 97 (14)

2. Primary Outcome: Contracture of Scar Surface Area (Percentage of Original Area)
Description: Contracture of Scar Surface Area 1 year post grafting: The surface area of the skin graft cm^2 at about one year after skin grafting will be compared to the size of the original skin graft at about one week after surgery.
Time Frame: 1 year post-grafting
Measure: Number; unit: percentage
Units Other Than Participants: skin burn area
Groups:
- Laser: Split person design
  Lidocaine Cream: Both sites will have lidocaine 4% topical anesthetic cream (Ferndale Laboratories, Ferndale MI) applied as thin layer and left for 30-45 minutes to minimize discomfort applied before laser treatment.
  Triamcinolone Acetonide Cream: Triamcinolone acetonide cream (Bristol-Myers Squibb, Princeton, NJ) at a concentration of 20mg/ml will be applied immediately after treatment to both laser and no-laser sites - as this is often reported and there is some speculation that this may be part of the reason improvement is noted.
  Fractional Ablative Laser: Applied to only site that is randomized to laser intervention
- No Laser: Split person design
  Lidocaine Cream: Both sites will have lidocaine 4% topical anesthetic cream (Ferndale Laboratories, Ferndale MI) applied as thin layer and left for 30-45 minutes to minimize discomfort applied before laser treatment.
  Triamcinolone Acetonide Cream: Triamcinolone acetonide cream (Bristol-Myers Squibb, Princeton, NJ) at a concentration of 20mg/ml will be applied immediately after treatment to both laser and no-laser sites - as this is often reported and there is some speculation that this may be part of the reason improvement is noted.
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 1 | 1
Number analyzed (skin burn area) | 1 | 1
percentage | 106 | 102

3. Secondary Outcome: Scar Roughness
Description: Scar Roughness at 9 weeks and 12 weeks post grafting: will be quantified using a mold/casting technique using Aquasil Ultra XLV dental impression material followed by mold imaging and quantitative analysis. A three-dimensional analysis of the molds will allow for measure of average roughness. The machine used will provide a digital read out which will then be averaged to obtain a mean value. This will allow for comparison between treated and control grafts at 90 days and one year.
Time Frame: 90 days post-grafting
Population: Data could not be collected. Unable to acquire molding due to COVID supply chain challenges.
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 0 | 0
Number analyzed (skin burn area) | 0 | 0

4. Secondary Outcome: Scar Roughness
Description: Scar Roughness 10-12 months post grafting: will be quantified using a mold/casting technique using Aquasil Ultra XLV dental impression material followed by mold imaging and quantitative analysis. A three-dimensional analysis of the molds will allow for measure of average roughness. The machine used will provide a digital read out that will then be averaged to obtain a mean value. This will allow for comparison between treated and control grafts at 90 days and one year.
Time Frame: 1 year post-grafting
Population: Data could not be collected. Unable to acquire molding due to COVID supply chain challenges.
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 0 | 0
Number analyzed (skin burn area) | 0 | 0

5. Secondary Outcome: Biomechanics Stiffness
Description: Biomechanics Stiffness 90 days post grafting: The BTC-2000 device uses a laser to measure skin deflection as negative atmospheric pressure is applied and this allows for quantification of the skin's mechanical properties (e.g. elasticity and stiffness). The device will provide a digital readout that will be averaged to obtain a mean value.
Time Frame: 90 days post-grafting
Measure: Mean (Standard Deviation); unit: kPa
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 8 | 8
Number analyzed (skin burn area) | 8 | 8
kPa | 206 (143) | 231 (187)

6. Secondary Outcome: Biomechanics Stiffness
Description: Biomechanics Stiffness 10-12 months post grafting: The BTC-2000 device uses a laser to measure skin deflection as negative atmospheric pressure is applied and this allows for quantification of the skin's mechanical properties (e.g. elasticity and stiffness). The device will provide a digital readout that will be averaged to obtain a mean value.
Time Frame: 1 year post-grafting
Measure: Mean (Standard Deviation); unit: kPa
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 1 | 1
Number analyzed (skin burn area) | 1 | 1
kPa | 283 (69) | 301 (48)

7. Secondary Outcome: Biomechanics Elasticity
Description: Elasticity will be quantified using a BTC-2000, a high resolution Target Laser and negative pressure transducer. The BTC-2000 device uses a laser to measure skin deflection as negative atmospheric pressure is applied and this allows for quantification of the skin's mechanical properties (e.g. elasticity and stiffness). The device will provide a digital readout that will be averaged to obtain a mean value.
Time Frame: 90 days post-grafting
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 8 | 8
Number analyzed (skin burn area) | 8 | 8
millimeters | 0.87 (0.52) | 0.66 (0.31)

8. Secondary Outcome: Biomechanics Elasticity
Description: as for outcome 7
Time Frame: 1 year post-grafting
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 1 | 1
Number analyzed (skin burn area) | 1 | 1
millimeters | 0.71 (0.28) | 0.71 (0.28)

9. Secondary Outcome: Erythema Index
Description: Erythema will be measured using a Mexameter that will accurately measure even small changes in erythema levels, then provide a digital read out from which an average mean can be obtained. The erythema levels are measured on a scale ranging from 0 to around 999. This index reflects the redness of the skin, which can be an indicator of various skin conditions or reactions. Higher index indicates a scar that is more red.
Time Frame: 90 days post-grafting
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 8 | 9
Number analyzed (skin burn area) | 8 | 9
score on a scale | 379 (117) | 360 (101)

10. Secondary Outcome: Erythema Index
Description: as for outcome 9
Time Frame: 1 year post-grafting
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 1 | 1
Number analyzed (skin burn area) | 1 | 1
score on a scale | 425 (35) | 384 (34)

11. Secondary Outcome: Vancouver Scar Scale (VSS)
Description: Scar-rating scale that objectively evaluates scar properties to include the following: Vascularity: Normal = 0, Pink=1, Red = 2, Purple = 3; Pigmentation: Normal= 0, Hypopigmentation= 1, Hyperpigmentation= 2; Pliability: Normal= 0, Supple =1, Yielding= 2, Firm= 3, Ropes= 4, Contracture= 5; Height: Flat= 0, <2mm=1, 2-5mm=2, >5mm=3; Lowest possible score= 0 and Highest Score possible = 13. Higher results denotes worse outcomes.
Time Frame: 90 days post-grafting
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 4 | 4
Number analyzed (skin burn area) | 4 | 4
score on a scale | 4.7 (1.0) | 4.7 (1.0)

12. Secondary Outcome: Vancouver Scar Scale (VSS)
Description: as for outcome 11
Time Frame: 1 year post-grafting
Measure: Number; unit: score on a scale
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 1 | 1
Number analyzed (skin burn area) | 1 | 1
score on a scale | 5 | 5

13. Secondary Outcome: Patient and Observer Scar Assessment Scale (POSAS)--Patient
Description: Subjective scar scale for the patient that measures perception of scar height, pliability, pigmentation, vascularization, and relief. Survey consists of seven questions with total score ranging from 7-70. The higher the score the worse the scar.
Time Frame: 90 days post-grafting
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 8 | 8
Number analyzed (skin burn area) | 8 | 8
score on a scale | 32 (5.4) | 36 (16)

14. Secondary Outcome: Patient and Observer Scar Assessment Scale (POSAS)--Observer
Description: Subjective scar scale for the observer measures perception of scar height, pliability, pigmentation, vascularization, and relief. Survey consists of six questions. Total score range 6-60. The higher the score the worse the scar.
Time Frame: 90 days post-grafting
Measure: Number; unit: score on a scale
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 1 | 1
Number analyzed (skin burn area) | 1 | 1
score on a scale | 19 | 18

15. Secondary Outcome: Patient and Observer Scar Assessment Scale (POSAS)--Patient
Description: as for outcome 13
Time Frame: 1 year post-grafting
Measure: Number; unit: score on a scale
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 1 | 1
Number analyzed (skin burn area) | 1 | 1
score on a scale | 19 | 19

16. Secondary Outcome: Patient and Observer Scar Assessment Scale (POSAS)--Observer
Description: as for outcome 14
Time Frame: 1 year post-grafting
Measure: Number; unit: score on a scale
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 1 | 1
Number analyzed (skin burn area) | 1 | 1
score on a scale | 13 | 14

17. Secondary Outcome: Patient-Reported Satisfaction
Description: Subjective measurement of patient satisfaction of outcome based on a 0-10 Likert scale with 10 being the best outcome.
Time Frame: 90 days post-grafting
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 8 | 8
Number analyzed (skin burn area) | 8 | 8
score on a scale | 5.25 (1.5) | 5.75 (1.89)

18. Secondary Outcome: Patient-Reported Satisfaction
Description: Subjective measurement of patient satisfaction of outcome based on a 0-10 Likert scale with 10 being the best outcome.
Time Frame: 1 year post-grafting
Measure: Number; unit: score on a scale
Units Other Than Participants: skin burn area
Arm/Group | Laser | No Laser
Number analyzed (Participants) | 1 | 1
Number analyzed (skin burn area) | 1 | 1
score on a scale | 3 | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Laser | No Laser
All-Cause Mortality (participants affected / at risk) | 1/9 | 1/9
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser (N=9) | No Laser (N=9)
death (Cardiac disorders) | 1 (1) | 1 (1) — cardiovascular embarrassment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT04176705/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT04176705/ICF_000.pdf